CLINICAL TRIAL: NCT01097239
Title: A Phase I/II Feasibility/Efficacy Study of HIFU in Otherwise Untreatable Pelvic Rectal Cancer
Brief Title: Examining the Role of Transrectal High Intensity Focused Ultrasound (HIFU) in Rectal Pelvic Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Failure to recruit.
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 09/H0808/43
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Rectal Cancer; Ovarian Cancer; Endometrial Cancer; Vaginal Cancer; Cervical Cancer
Keywords: High Intensity Focused Ultrasound; HIFU; Rectal Cancer; Sonablate 500; Transrectal
MeSH Terms: conditions — Rectal Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Vaginal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Intensity Focused Ultrasound (Experimental): Transrectal High Intensity Focused Ultrasound (HIFU) treatment of the PelvicTumour
  Interventions: Device: Sonablate 500 (High Intensity Focused Ultrasound (HIFU))

INTERVENTIONS:
Device: Sonablate 500 (High Intensity Focused Ultrasound (HIFU)) — High Intensity Focused Ultrasound (HIFU) Delivered by the Sonablate 500 Transrectal Device
  Other Names: Sonablate 500; HIFU

SUMMARY:
This is a single centre pilot trial to establish the feasibility and role of endoluminal HIFU in patients with locally advanced cancer within the pelvis that is either primary or recurrent and with all available current therapy inappropriate and/or exhausted.

The aim is to make a preliminary assessment of efficacy & dosage for evaluation in a randomised controlled trial. Whilst efficacy data are limited in a small feasibility study; radiological, biochemical and histopathological analysis of the patient and patient specimens, along with quality of life questionnaires (QoL), will be used to provide preliminary measures of efficacy in this patient cohort.

These analyses will allow examination of the biochemical, metabolomic and histological changes associated with HIFU treatment in cancer within the pelvis.

DETAILED DESCRIPTION:
CURRENT TREATMENT OF LOCALLY ADVANCED PELVIC CANCER Colorectal cancer This is a common condition with about 40,000 new cases a year in the United Kingdom. The optimal multimodality management of stage III & IV rectal cancer remains an increasing challenge. There is a high risk of local recurrence and poor survival has been reported for patients treated by surgery alone. About 20% of patients may present with locally advanced tumours, which are partially or totally fixed (T3/T4). Until recently there have been no widely accepted and validated methods of defining preoperatively either locally advanced rectal cancer or unresectable disease. The use of pre-operative pelvic magnetic resonance imaging (MRI) to predict the likelihood of achieving an R0 resection (Beets-Tan et al 2001, Brown et al 2003) has resulted in improved selection. Pre-operative chemoradiotherapy can downstage locally advanced tumours, and result in higher resection rates being achieved with reduced risk of local recurrence (Bosset et al 1993, Rich et al 1995).

Gynaecological cancers Treating other advanced pelvic malignancies including vaginal, ovarian, endometrial and cervical cancers is similarly challenging. Disease recurrence at the site of surgical resection or adjacent lymph nodes can also preclude further curative options, due to chemotherapy resistance, reaching maximum safe radiotherapy limits or unsuitable surgical options.

It is proposed that High Intensity Focused Ultrasound (HIFU) may become another modality of treatment in locally advanced or unresectable pelvic disease.

RATIONALE FOR PERFORMING THE STUDY Colorectal cancer This is the third most common cause of cancer and cancer death in both men and women (40,000 cases and just under 16 000 deaths per year in the UK). Worldwide, there are approximately 1 million cases and 500 000 deaths per annum. Primary treatment is usually surgical with, in appropriate cases, adjuvant or neo-adjuvant therapy currently including radiotherapy, cytotoxic chemotherapy or a combination. Unfortunately, the overall survival of locally advanced disease is at best 50%. Many patients who have residual, refractory or recurrent rectal cancer experience serious morbidity from local tumour invading and destroying adjacent tissues including bone, nerves (sacrum), bladder and the skin. These interfere severely with normal daily activities, especially bowel function and cause great distress in terms of pain, with many patients requiring permanent palliative colostomies.

Gynaecological cancers Other advanced pelvic malignancies can be equally problematic to manage successfully. Annually in the UK, approximately 250 vaginal cancer, 7000 ovarian cancer, 8000 endometrial cancer and 3000 cervical cancer diagnoses are made, with some being incurable at the time of presentation. Treatment options include surgery, hormonal therapy, chemotherapy, radiotherapy or a combination, although palliative patients can often be left with debilitating symptoms including severe pain and fistula formation, compromising their quality of life.

High Intensity Focused Ultrasound (HIFU) is a method of accurately delivering ablative ultrasound (US) generated high temperatures non-invasively or endo-luminally focused to specific areas in the body using imaging (ultrasound or MR) guidance. Intracavitary or endo-luminal (also called transrectal) HIFU has been appraised by the National Institute for Clinical Excellence (NICE) in the treatment of prostate cancer. It is currently used for primary prostate cancer; there is also evidence it may be effective in treating post-radiotherapy prostate cancer recurrence. Short and medium term data demonstrate that HIFU may be equivalent to some current prostate cancer therapies but with reduced morbidity and length of stay. As the prostate and rectum are adjacent there is now a natural evolution to translate the success in prostate to the adjacent rectum/other pelvic structures.

There is a large unmet clinical need for new treatments for patients with residual or progressing local pelvic cancer (such as rectal in origin as well as other pelvic malignancies) in whom all current therapies are exhausted. Intracavitary HIFU offers such a therapy.

An initial cohort of 20 patients will be offered intracavitary HIFU using the Sonablate 500 (Sonacare Medical, Charlotte, NC, USA) intra-luminal device (at different, escalating energy doses) under general anaesthetic with monitoring for toxicity and ablative efficacy using pre and post-treatment Imaging.

As none of the intracavitary devices have yet been used in rectal, vaginal, ovarian, endometrial, cervical or pelvic lymph node tumours directly (but have been used in the rectum to treat prostate cancer), it is important that to gauge the levels of energy and resultant cancer tissue destruction from a variety of different treatment energies. In this manner, the first phase of this trial is equivalent to the 'dose escalation' phase of a drug trial.

Once the optimum energy levels, safety and treatment protocol are known, a further 30 patients will be treated in Phase II. Patients will undergo MR Imaging pre- and post-treatment to objectively assess the tumour and will complete quality of life questionnaires, pain scores, and functional questionnaires. Survival data will be documented. Post-treatment imaging will be performed at between 3-4 weeks, as within this time frame the ablative effect (a necrotic area) as seen in prostate cancer treated by HIFU, will become clearer providing useful data for the Phase I element.

The trial will run in two stages: the end of the first phase (for regulatory requirements) is defined as 30 days from the date that the last patient has completed trial therapy. The non-interventional follow-up stage will then commence in which patients are followed up for a minimum of 6 months or death.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven rectal, vaginal, ovarian, endometrial or cervical cancer (tumour <15cm from anal/vaginal verge)
* Lymph node(s) accessible by HIFU for which the primary clinical team advise intervention
* Partially fixed/unresectable disease and locally advanced disease (T3/T4)
* Patient considered to be unsuitable for or have exhausted all currently available therapies
* WHO Performance Status 0-2
* Fit for general anaesthetic and HIFU
* Not pregnant
* No other serious uncontrolled concomitant illness likely to interfere with treatment or assessment
* Written informed consent for treatment

Exclusion Criteria:

* WHO performance status of 3 or more
* Uncontrolled cardiac, respiratory or other disease, or any serious medical or psychiatric disorder that would preclude anaesthetic or informed consent
* Pelvic sepsis
* Currently enrolled in any other treatment trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Quality of life scores (EORTC QLQ-C30 and/or EORTC QLQ-CR38, EORTC QLQ-CX24, EORTC QLQ-EN24 or EORTC QLQ-OV24) | Within the first 30, 60 and 90 days after HIFU
  Validated Quality of Life Questionnaire

SECONDARY OUTCOMES:
Pain relief visual analogue scale | Within the first 30, 60 and 90 days after HIFU
Tumour marker changes (CEA and CA19.9) | Within the first 30, 60 and 90 days after HIFU

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Abel, ChM FRCS(Lon) FRCS(Ed), Principal Investigator — Imperial College London; Leonardo Monzon, BSc MBBS MRCS(Eng), Study Chair — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust (Hammersmith Hospital), London, England, United Kingdom

REFERENCES:
- [Background] Thuroff S, Chaussy C, Vallancien G, Wieland W, Kiel HJ, Le Duc A, Desgrandchamps F, De La Rosette JJ, Gelet A. High-intensity focused ultrasound and localized prostate cancer: efficacy results from the European multicentric study. J Endourol. 2003 Oct;17(8):673-7. doi: 10.1089/089277903322518699. PMID 14622488
- [Background] Hill CR, ter Haar GR. Review article: high intensity focused ultrasound--potential for cancer treatment. Br J Radiol. 1995 Dec;68(816):1296-1303. doi: 10.1259/0007-1285-68-816-1296. PMID 8777589
- [Background] Thuroff S, Chaussy C. High-intensity focused ultrasound: complications and adverse events. Mol Urol. 2000 Fall;4(3):183-7;discussion 189. PMID 11062373
- [Background] Visioli AG, Rivens IH, ter Haar GR, Horwich A, Huddart RA, Moskovic E, Padhani A, Glees J. Preliminary results of a phase I dose escalation clinical trial using focused ultrasound in the treatment of localised tumours. Eur J Ultrasound. 1999 Mar;9(1):11-8. doi: 10.1016/s0929-8266(99)00009-9. PMID 10099162
- [Background] Wu F, Chen WZ, Bai J, Zou JZ, Wang ZL, Zhu H, Wang ZB. Pathological changes in human malignant carcinoma treated with high-intensity focused ultrasound. Ultrasound Med Biol. 2001 Aug;27(8):1099-106. doi: 10.1016/s0301-5629(01)00389-1. PMID 11527596
- [Background] Wu F, Wang ZB, Chen WZ, Bai J, Zhu H, Qiao TY. Preliminary experience using high intensity focused ultrasound for the treatment of patients with advanced stage renal malignancy. J Urol. 2003 Dec;170(6 Pt 1):2237-40. doi: 10.1097/01.ju.0000097123.34790.70. PMID 14634387
- [Background] Stewart EA, Gedroyc WM, Tempany CM, Quade BJ, Inbar Y, Ehrenstein T, Shushan A, Hindley JT, Goldin RD, David M, Sklair M, Rabinovici J. Focused ultrasound treatment of uterine fibroid tumors: safety and feasibility of a noninvasive thermoablative technique. Am J Obstet Gynecol. 2003 Jul;189(1):48-54. doi: 10.1067/mob.2003.345. PMID 12861137
- [Background] Blana A, Walter B, Rogenhofer S, Wieland WF. High-intensity focused ultrasound for the treatment of localized prostate cancer: 5-year experience. Urology. 2004 Feb;63(2):297-300. doi: 10.1016/j.urology.2003.09.020. PMID 14972475
- [Background] Gelet A, Chapelon JY, Poissonnier L, Bouvier R, Rouviere O, Curiel L, Janier M, Vallancien G. Local recurrence of prostate cancer after external beam radiotherapy: early experience of salvage therapy using high-intensity focused ultrasonography. Urology. 2004 Apr;63(4):625-9. doi: 10.1016/j.urology.2004.01.002. PMID 15072864
- [Background] Wu F, Wang ZB, Cao YD, Chen WZ, Bai J, Zou JZ, Zhu H. A randomised clinical trial of high-intensity focused ultrasound ablation for the treatment of patients with localised breast cancer. Br J Cancer. 2003 Dec 15;89(12):2227-33. doi: 10.1038/sj.bjc.6601411. PMID 14676799
- [Background] Moore WE, Lopez RM, Matthews DE, Sheets PW, Etchison MR, Hurwitz AS, Chalian AA, Fry FJ, Vane DW, Grosfeld JL. Evaluation of high-intensity therapeutic ultrasound irradiation in the treatment of experimental hepatoma. J Pediatr Surg. 1989 Jan;24(1):30-3; discussion 33. doi: 10.1016/s0022-3468(89)80295-7. PMID 2723989
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Beets-Tan RG, Beets GL, Vliegen RF, Kessels AG, Van Boven H, De Bruine A, von Meyenfeldt MF, Baeten CG, van Engelshoven JM. Accuracy of magnetic resonance imaging in prediction of tumour-free resection margin in rectal cancer surgery. Lancet. 2001 Feb 17;357(9255):497-504. doi: 10.1016/s0140-6736(00)04040-x. PMID 11229667
- [Background] Quirke P, Durdey P, Dixon MF, Williams NS. Local recurrence of rectal adenocarcinoma due to inadequate surgical resection. Histopathological study of lateral tumour spread and surgical excision. Lancet. 1986 Nov 1;2(8514):996-9. doi: 10.1016/s0140-6736(86)92612-7. PMID 2430152
- [Background] Fazio VW, Tekkis PP, Remzi F, Lavery IC. Assessment of operative risk in colorectal cancer surgery: the Cleveland Clinic Foundation colorectal cancer model. Dis Colon Rectum. 2004 Dec;47(12):2015-24. doi: 10.1007/s10350-004-0704-y. PMID 15657649
- [Background] Buess G, Mentges B, Manncke K, Starlinger M, Becker HD. Technique and results of transanal endoscopic microsurgery in early rectal cancer. Am J Surg. 1992 Jan;163(1):63-9; discussion 69-70. doi: 10.1016/0002-9610(92)90254-o. PMID 1733375
- See also: Related Info — http://www.ukhifu.co.uk/
- See also: Related Info — http://www3.imperial.ac.uk/
- See also: Related Info — http://www.cancerhelp.org.uk/about-cancer/cancer-questions/high-intensity-focused-ultrasound